CLINICAL TRIAL: NCT01693601
Title: Panobinostat and Ruxolitinib In MyElofibrosis (PRIME STUDY) - Phase I/II Study of Combination Oral JAK2 Tyrosine Kinase Inhibitor (JAK2-TKI) and Histone Deacetylase Inhibitor (HDACI) Therapy in Patients With Myelofibrosis
Brief Title: Panobinostat and Ruxolitinib In MyElofibrosis (PRIME Trial)
Acronym: PRIME
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: John Mascarenhas (Other)
Responsible Party: Sponsor-Investigator, John Mascarenhas, Associate Professor of Medicine, Hematology and Medical Oncology, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GCO 12-1225
Record Dates: First submitted 2012-09-14; First posted 2012-09-26 (Estimated); Results first posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Myelofibrosis
Keywords: Myelofibrosis; Panobinostat; Ruxolitinib
MeSH Terms: conditions — Primary Myelofibrosis | interventions — Panobinostat; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Panobinostat and Ruxolitinib (Experimental): Combination of Panobinostat and Ruxolitinib
  Interventions: Drug: Panobinostat; Drug: Ruxolitinib

INTERVENTIONS:
Drug: Panobinostat — PO TIW QOW or PO TIW QW
  Other Names: LBH589
Drug: Ruxolitinib — PO BID x 28 days
  Other Names: INCB424, Jakafi

SUMMARY:
This is a single-center, single arm, dose finding study to assess safety and tolerability of the oral combination of Panobinostat and Ruxolitinib in patients with myelofibrosis (MF) in chronic and accelerated phase.

DETAILED DESCRIPTION:
Phase I/II open label, single institution, combination therapy trial of induction Ruxolitinib followed by combination with Panobinostat in dose escalation cohorts with a primary endpoint of determining the safety and tolerability of combination therapy in patients with myelofibrosis (MF) in chronic and accelerated phase. A 3+3standard dose escalation scheme will be employed and the occurrence of dose limiting toxicities (DLTs) will be captured and the occurrence of such events will determine dose cohort escalation by predetermined and established rules. In addition to establishing the DLTs, maximally tolerated dose (MTD), and recommended phase II dose (RPTD) in the phase I portion of this trial, exploratory biomarkers will be evaluated within phase I as well. Pharmacodynamics and exploratory genetic and epigenetic biomarkers will be explored as predictors of response to therapy. The RPTD cohort will be expanded to incorporate a total of 22 patients, including 6 from phase I, in order to assess clinical response as assessed by International Working Group for Myelofibrosis Research and Treatment (IWG-MRT) as a primary endpoint for the phase II portion of this trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥ 18 years old
* Ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
* Intermediate-2 and higher by IWG-MRT Post PV/ET MF and PMF patients either in

  1. Chronic Phase (MF-CP)
  2. Accelerated Phase (MF-AP)
* Patients must meet the following laboratory criteria:

  1. ANC ≥ .750 x 109/L
  2. Platelets ≥ 75 x 109/L
  3. Creatinine ≤ 1.5 x ULN,
  4. AST and ALT ≤ 2.5 x ULN
  5. Serum bilirubin ≤ 1.5 x ULN (unless Gilbert's syndrome and evidence of hemolysis)
  6. Serum potassium ≥ LLN
  7. Total serum calcium [corrected for serum albumin] or ionized calcium ≥LLN,
  8. Serum magnesium ≥ LLN
  9. Serum phosphorus ≥ LLN
  10. Free T4 within normal limits
* ECOG Performance Status of ≤ 3
* Any prior therapy with JAK2-TKI, hypomethylating agents, HDACI, mTORi, or iMiDs is allowed as long as it is greater than 3 weeks since last dose of administration and in the case of a JAK2-TKI or HDACI that discontinuation was not due to non-hematologic drug toxicity. An exception to this criteria are patients currently on at least 10mg BID of ruxolitinib for greater than 3 months and who have not shown an optimal response (i.e. without 50% reduction in palpable splenomegaly or 50% reduction in symptom burden). With a reduction of ruxolitinib to 10mg BID these patients may enter onto the study without stopping ruxolitinib

Exclusion Criteria:

* Patients who will need valproic acid for any medical condition during the study or within 5 days prior to first PANOBINOSTAT treatment.
* Impaired cardiac function or clinically significant cardiac diseases, including any one of the following:

  1. With permanent cardiac pacemaker
  2. Resting bradycardia defined as <50 beats per minute
  3. QTcF >450 msec on screening ECG
  4. Complete Left bundle branch block, bifascicular block
  5. Any clinically significant ST segment and/or T-wave abnormalities
  6. Presence of unstable atrial fibrillation (ventricular response rate >100 bpm). Patients with stable atrial fibrillation can be enrolled provided they do not meet other cardiac exclusion criteria.
  7. Symptomatic congestive heart failure (NYHA class III-IV)
* Impairment of GI function or GI disease that may significantly alter the absorption of PANOBINOSTAT or RUXOLITINIB
* Other concurrent severe and/or uncontrolled medical conditions (e.g., uncontrolled diabetes or active or uncontrolled infection) including abnormal laboratory values, that could cause unacceptable safety risks or compromise compliance with the protocol
* Patients using medications that have a relative risk of prolonging the QT interval or inducing torsade de pointes if treatment cannot be discontinued or switched to a different medication prior to starting study drug
* Concomitant use of CYP3A4 inhibitors
* Patients who have received targeted agents within 2 weeks or within 5 half-lives of the agent and active metabolites (whichever is longer) and who have not recovered from side effects of those therapies.
* Chemotherapy within 3 weeks prior to screening are excluded (other than hydroxyurea at stable doses and will be discontinued 24 hours prior to starting study drug).
* Patients with an active bleeding tendency or are receiving any treatment with therapeutic doses of sodium warfarin (Coumadin®) or coumadin derivatives. Patients will be allowed to enter study on aspirin at doses of 81mg/d.
* Patients who have undergone major surgery ≤ 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* Women who are pregnant or breast-feeding or women of childbearing potential (WOCBP) not using an effective method of birth control. WOCBP are defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months). Women of childbearing potential must have a negative serum pregnancy test within 24hrs of receiving the first dose of study medication.
* Male patients whose sexual partners are WOCBP not using effective birth control
* Patients with a prior malignancy within the last 5 years (except for basal or squamous cell carcinoma, or in situ cancer of the cervix)
* Disease associated with secondary MF such as metastatic carcinoma, lymphoma, myelodysplasia, hairy cell leukemia, mast cell disease or acute leukemia (including M7 disease or acute panmyelosis with MF)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-01; Primary Completion 2018-05-18 (Actual); Study Completion 2018-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Mascarenhas, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Result] Mascarenhas J, Marcellino BK, Lu M, Kremyanskaya M, Fabris F, Sandy L, Mehrotra M, Houldsworth J, Najfeld V, El Jamal S, Petersen B, Moshier E, Hoffman R. A phase I study of panobinostat and ruxolitinib in patients with primary myelofibrosis (PMF) and post--polycythemia vera/essential thrombocythemia myelofibrosis (post--PV/ET MF). Leuk Res. 2020 Jan;88:106272. doi: 10.1016/j.leukres.2019.106272. Epub 2019 Nov 16. PMID 31778911

RESULTS

PARTICIPANT FLOW:
Groups:
- Panobinostat and Ruxolitinib Cohort 1: Combination of Panobinostat 10mg and Ruxolitinib 10mg
- Panobinostat and Ruxolitinib Cohort 2: Combination of Panobinostat 10mg and Ruxolitinib 15mg
- Panobinostat and Ruxolitinib Cohort 3: Combination of Panobinostat 10mg and Ruxolitinib 20mg
- Panobinostat and Ruxolitinib Cohort 4: Combination of Panobinostat 15mg and Ruxolitinib 15mg
Period: Cohort 1
Arm/Group | Panobinostat and Ruxolitinib Cohort 1 | Panobinostat and Ruxolitinib Cohort 2 | Panobinostat and Ruxolitinib Cohort 3 | Panobinostat and Ruxolitinib Cohort 4
Started | 3 | 0 | 0 | 0
Completed | 3 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Cohort 2
Arm/Group | Panobinostat and Ruxolitinib Cohort 1 | Panobinostat and Ruxolitinib Cohort 2 | Panobinostat and Ruxolitinib Cohort 3 | Panobinostat and Ruxolitinib Cohort 4
Started | 0 | 6 | 0 | 0
Completed | 0 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Cohort 3
Arm/Group | Panobinostat and Ruxolitinib Cohort 1 | Panobinostat and Ruxolitinib Cohort 2 | Panobinostat and Ruxolitinib Cohort 3 | Panobinostat and Ruxolitinib Cohort 4
Started | 0 | 0 | 3 | 0
Completed | 0 | 0 | 3 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Cohort 4
Arm/Group | Panobinostat and Ruxolitinib Cohort 1 | Panobinostat and Ruxolitinib Cohort 2 | Panobinostat and Ruxolitinib Cohort 3 | Panobinostat and Ruxolitinib Cohort 4
Started | 0 | 0 | 0 | 3
Completed | 0 | 0 | 0 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Panobinostat and Ruxolitinib Cohort 1 | Panobinostat and Ruxolitinib Cohort 2 | Panobinostat and Ruxolitinib Cohort 3 | Panobinostat and Ruxolitinib Cohort 4 | Total
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 15
Age, Continuous [Median (Full Range); unit: years] | 60 [53 to 74] | 61 [52 to 78] | 69 [46 to 78] | 64 [64 to 66] | 64 [46 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 1 | 4
  Male | 2 | 5 | 2 | 2 | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Disease subtype [Count of Participants; unit: Participants]
  Primary myelofibrosis (PMF) | 1 | 3 | 1 | 1 | 6
  Post essential thrombocythemia PET-MF | 2 | 3 | 1 | 1 | 7
  Post polycythemia vera PPV-MF | 0 | 0 | 1 | 1 | 2
DIPSS Score [Count of Participants; unit: Participants] — Dynamic International Prognostic Scoring System (DIPSS) for PMF uses five risk factors to predict survival: age older than 65 years, hemoglobin lower than 10 g/dL, leukocytes higher than 25 × 10(9)/L, circulating blasts ≥ 1%, and constitutional symptoms. Total score range from 0-6, with higher score indicating more risk and lower median year survival.
  Participants
    low (score 0) | 1 | 0 | 0 | 0 | 1
    intermediate-1 (score 1 or 2) | 0 | 2 | 3 | 1 | 6
    intermediate-2 (score 3 or 4) | 2 | 4 | 0 | 2 | 8
JAK2^V617F positive [Count of Participants; unit: Participants] | 3 | 4 | 2 | 1 | 10
Cytogenetics [Count of Participants; unit: Participants]
  Unfavorable Karyotype | 0 | 2 | 0 | 0 | 2
  Not Unfavorable Karyotype | 1 | 4 | 3 | 3 | 11
  Not available | 2 | 0 | 0 | 0 | 2
Prior Myelofibrous (MF) Directed Therapy [Count of Participants; unit: Participants] | 2 | 6 | 2 | 1 | 11
Ruxolitinib Naive [Count of Participants; unit: Participants] | 3 | 3 | 2 | 2 | 10
Prior No. Therapies [Median (Full Range); unit: therapies] | 1 [0 to 3] | 1.5 [1 to 4] | 2 [0 to 4] | 0 [0 to 3] | 1 [0 to 4]
Red Blood Cell (RBC) Transfusion Dependent [Count of Participants; unit: Participants] — each cycle is 28 days
  Participants
    Screening | 1 | 1 | 0 | 0 | 2
    Baseline - Cycle 1, Day 1 (C1D1) Rux +Pano | 1 | 1 | 1 | 0 | 3
White Blood Cell (WBC) [Median (Full Range); unit: 10^3 cells/µl]
  Screening | 11.3 [4 to 13.4] | 9.8 [2.8 to 32.9] | 9.8 [4.3 to 16.7] | 34.3 [12.5 to 39.3] | 12.5 [2.8 to 39.3]
  Baseline, C1D1 | 5.1 [2.9 to 6.2] | 7 [4.3 to 34.6] | 6 [5.3 to 22.4] | 25.9 [11.9 to 30.4] | 6.8 [2.9 to 34.6]
Hemoglobin (Hb) [Median (Full Range); unit: g/DL]
  Screening | 9.1 [8.7 to 12] | 9.7 [8.3 to 11.9] | 10.5 [8.6 to 11] | 11.2 [9.8 to 12.8] | 9.8 [8.3 to 12.8]
  Baseline, C1D1 | 8.4 [7.9 to 11.2] | 10.75 [6.9 to 12.2] | 10.1 [9.4 to 10.4] | 11.7 [9.9 to 13] | 10.4 [6.9 to 13]
Platelet (PLT) [Median (Full Range); unit: 10^3 cells/µl]
  Screening | 495 [159 to 672] | 276 [95 to 463] | 584 [183 to 584] | 377 [206 to 407] | 347 [95 to 672]
  Baseline, C1D1 | 131 [67 to 307] | 192.5 [82 to 729] | 166 [139 to 621] | 253 [160 to 379] | 188 [67 to 729]
Palpable Spleen [Count of Participants; unit: Participants]
  Screening | 3 | 5 | 2 | 3 | 13
  Baseline, C1D1 | 2 | 5 | 1 | 3 | 11
Palpable Spleen Length [Median (Full Range); unit: cm]
  Screening | 6 [2 to 14] | 12.5 [0 to 18] | 10 [0 to 14] | 15 [13 to 17] | 13 [0 to 18]
  Baseline, C1D1 | 6 [0 to 10] | 11 [0 to 16] | 0 [0 to 15] | 11 [10 to 15] | 10 [0 to 16]
MRI Spleen Volume [Median (Full Range); unit: cm^3] | 1190 [874 to 2655] | 2154.5 [1573 to 3950] | 2425 [346 to 2773] | 1982 [1971 to 2544] | 2077 [346 to 3950]

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients That Achieve Stable Disease or Clinical Improvement
Description: Number of patients that have either stable disease or clinical improvement treatment response as defined by the International Working Group for Myelofibrosis Research and Treatment (IWG-MRT).
  Stable disease (SD) - response that is not complete remission, partial remission, clinical improvement, anemia response, spleen response, symptoms response, or progressive disease.
  Clinical improvement (CI) - a response in anemia, splenomegaly, or MF-SB that is not associated with progressive splenomegaly or increase in severity of anemia, thrombocytopenia, or neutropenia.
Time Frame: at least 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Panobinostat and Ruxolitinib Cohort 1 | Panobinostat and Ruxolitinib Cohort 2 | Panobinostat and Ruxolitinib Cohort 3 | Panobinostat and Ruxolitinib Cohort 4
Number analyzed (Participants) | 3 | 6 | 3 | 3
Participants
  Stable disease | 3 | 4 | 1 | 3
  Clinical Improvement | 0 | 1 | 2 | 0
  No response evaluated | 0 | 1 | 0 | 0

2. Primary Outcome: Number of Participants Who Experienced Dose-Limiting (DLTs)
Description: Panobinostat related adverse events requiring dose reduction or discontinuing prior to Cycle 6, Day 29 (C6D29)
Time Frame: up to cycle 6, day 29
Measure: Count of Participants; unit: Participants
Arm/Group | Panobinostat and Ruxolitinib Cohort 1 | Panobinostat and Ruxolitinib Cohort 2 | Panobinostat and Ruxolitinib Cohort 3 | Panobinostat and Ruxolitinib Cohort 4
Number analyzed (Participants) | 3 | 6 | 3 | 3
Participants
  requiring Panaobinostat dose reduction | 1 | 0 | 3 | 1
  Discontinuing Panobinostat | 0 | 2 | 0 | 0

3. Secondary Outcome: Percent Change in Spleen Volume
Description: Percent change in spleen volume at C6D29 as compared to baseline
Time Frame: Baseline and Cycle 6, Day 29
Population: One participant did not return for C6,D29 visit
Measure: Median (Full Range); unit: percent change
Arm/Group | Panobinostat and Ruxolitinib Cohort 1 | Panobinostat and Ruxolitinib Cohort 2 | Panobinostat and Ruxolitinib Cohort 3 | Panobinostat and Ruxolitinib Cohort 4
Number analyzed (Participants) | 3 | 5 | 3 | 3
percent change | -41 [-44 to -8] | -8 [-61 to 25] | -40 [-59 to 4] | -17 [-29 to -15]

4. Secondary Outcome: Percent Change in Spleen Size for Responders and Non-responders
Description: Percent change in spleen length size by palpation at cycle 6, day 29 (C6D29) from baseline
Time Frame: Cycle 6, Day 29
Measure: Median (Full Range); unit: percent change
Groups:
- Responders: Responders are those participants who were listed as Clinical Improvement (CI) as assessed by the IWG Response
- Non-Responders: Non-Responders are those participants who were listed as Stable Disease (SD) as assessed by the IWG Response. Participant who had no response evaluated also included in this group.
Arm/Group | Responders | Non-Responders
Number analyzed (Participants) | 3 | 12
percent change | -100 [-100 to -14] | -29 [-100 to 0]

5. Secondary Outcome: Percent Change in Spleen Length
Description: Percent change in spleen length at C6D29
Time Frame: Cycle 6, Day 29
Population: One participant did not return for C6,D29 visit
Measure: Median (Full Range); unit: percent change
Arm/Group | Panobinostat and Ruxolitinib Cohort 1 | Panobinostat and Ruxolitinib Cohort 2 | Panobinostat and Ruxolitinib Cohort 3 | Panobinostat and Ruxolitinib Cohort 4
Number analyzed (Participants) | 3 | 5 | 3 | 3
percent change | -83 [-100 to -29] | -17 [-100 to 0] | -14 [-100 to 0] | -31 [-33 to -29]

6. Secondary Outcome: Number of Participants With Percent Change on Myeloproliferative Neoplasm Symptom Assessment Form (MPN-SAF)
Description: Symptom responders defined as having a percent change in MPN-SAF score from Screening/C1D1 to C6D29 of more than 50%.MPN-SAF is an 18-item instrument. Each item score 0-10 averaged, total scale from0-10, with higher score indicating more symptoms.
Time Frame: baseline, C1D1 and Cycle 6 Day 29
Population: C6D29 not available for one participant in cohort 2 and 2 participants in cohort 4
Measure: Count of Participants; unit: Participants
Arm/Group | Panobinostat and Ruxolitinib Cohort 1 | Panobinostat and Ruxolitinib Cohort 2 | Panobinostat and Ruxolitinib Cohort 3 | Panobinostat and Ruxolitinib Cohort 4
Number analyzed (Participants) | 3 | 5 | 3 | 1
Participants | 1 | 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Panobinostat and Ruxolitinib Cohort 1 | Panobinostat and Ruxolitinib Cohort 2 | Panobinostat and Ruxolitinib Cohort 3 | Panobinostat and Ruxolitinib Cohort 4
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/6 | 3/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panobinostat and Ruxolitinib Cohort 1 (N=3) | Panobinostat and Ruxolitinib Cohort 2 (N=6) | Panobinostat and Ruxolitinib Cohort 3 (N=3) | Panobinostat and Ruxolitinib Cohort 4 (N=3)
Anemia (Blood and lymphatic system disorders) | 1 | 2 | 2 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0
Night Sweats (General disorders) | 0 | 0 | 1 | 0
Oral Ulcers (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Ruxolitinib withdrawal (Product Issues) | 0 | 1 | 0 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Prostate ca in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Wound complication post surgery (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fever (General disorders) | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0
Supraventricula Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Bilateral PE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panobinostat and Ruxolitinib Cohort 1 (N=3) | Panobinostat and Ruxolitinib Cohort 2 (N=6) | Panobinostat and Ruxolitinib Cohort 3 (N=3) | Panobinostat and Ruxolitinib Cohort 4 (N=3)
Anemia (Blood and lymphatic system disorders) | 1 | 2 | 2 | 2
Upper Respiratory Infection (Infections and infestations) | 1 | 4 | 2 | 1
Diarrhea (Gastrointestinal disorders) | 3 | 3 | 2 | 2
Headache (Nervous system disorders) | 1 | 2 | 0 | 2
Vertigo (Ear and labyrinth disorders) | 1 | 2 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1 | 1
Abdominal bloating (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 2 | 0 | 1
Night Sweats (General disorders) | 1 | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Oral Ulcers (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Hypertension (Vascular disorders) | 1 | 2 | 1 | 0
Leg Cramps (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Taste changes (Nervous system disorders) | 0 | 3 | 1 | 1
Ankle Swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Chest Pain (Cardiac disorders) | 0 | 1 | 0 | 0
Edema (General disorders) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0
Fever (General disorders) | 0 | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 1
Spleen pain (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0
Weight Gain (Investigations) | 1 | 1 | 1 | 0
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0
Chills (General disorders) | 0 | 2 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 2 | 0 | 0 | 0
Frequent Urination (Renal and urinary disorders) | 0 | 0 | 0 | 0
Fungal Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Gastroesophageal Reflux (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hematoma (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Hematuria (Renal and urinary disorders) | 1 | 0 | 1 | 0
Leg Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rectal Bleeding (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Squamous Cell Lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0
Clavicular Protuberance (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin Rash/Infection (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Prostatitis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Bleeding (finger) (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Paresthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dysphagia (Nervous system disorders) | 0 | 0 | 3 | 0
Early Satiety (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Emotional lability (Psychiatric disorders) | 0 | 0 | 1 | 0
Folliculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Gum Bleeding (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Increased dental plaque (General disorders) | 0 | 1 | 0 | 0
Broken tooth (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Blockage of left medial canthus (Eye disorders) | 0 | 0 | 0 | 1
Blurry vision (Eye disorders) | 0 | 0 | 0 | 1
Baker's cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Bilirubin increased (Investigations) | 0 | 0 | 1 | 0
Creatinine increased (Investigations) | 0 | 1 | 0 | 0
Facial pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1
Eye itching (right) (Eye disorders) | 0 | 0 | 0 | 1
Grover's disease (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Muscle aches (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Nipple pain (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Nocturnal myoclonic jerks (General disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-19): https://cdn.clinicaltrials.gov/large-docs/01/NCT01693601/Prot_SAP_000.pdf